CLINICAL TRIAL: NCT00812903
Title: Neck Pain in Danish Military Pilots and Flight Crew - Environmental Factors With Influence on Performance (PH.D.-Project)
Brief Title: Neck Pain in Danish Military Pilots and Flight Crew
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Danish Defence (Unknown); Royal Danish Air Force (Unknown)
Responsible Party: Principal Investigator, Britt Lange, MD, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-20090005
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Neck Pain
Keywords: Neck; Pain; Exercise; Pilots; Crew
MeSH Terms: conditions — Neck Pain; Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control group
- Exercise (Experimental): Intervention group
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Training exercises chosen with background in knowledge of intelligent training
  Other Names: Training
  Arms: Exercise

SUMMARY:
The purpose of this study is to determine the prevalence of neck and shoulder pain in Danish fighter pilots, helicopter pilots and helicopter flight crew and to evaluate the effect of a 24 weeks exercise intervention for fighter pilots.

ELIGIBILITY:
Inclusion Criteria:

* Military fighter and helicopter pilots and crew
* Active flying 2006 or later

Exclusion Criteria:

* Pilots and crew not active since 2005 or earlier
* Pilots and crew with other nationality than Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Neck pain | 1 year
Compliance to training exercises | 1 year

SECONDARY OUTCOMES:
Muscle strength | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Sjoegaard, Professor, Study Director — University of Souther Denmark
Locations (1):
- Fighterwing Skrydstrup, Vojens, Denmark

REFERENCES:
- [Background] Jones JA, Hart SF, Baskin DS, Effenhauser R, Johnson SL, Novas MA, Jennings R, Davis J. Human and behavioral factors contributing to spine-based neurological cockpit injuries in pilots of high-performance aircraft: recommendations for management and prevention. Mil Med. 2000 Jan;165(1):6-12. PMID 10658420